CLINICAL TRIAL: NCT07002151
Title: Effect of Educational Kinesiology Program on Cognition, Manual Dexterity and Bimanual Coordination in Patients With Multiple Sclerosis
Brief Title: Educational Kinesiology Program's Effect on Cognition, Manual Dexterity and Bimanual Coordination in MS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mona abo-elabbas ahmed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: effect of EKP on cognition
Record Dates: First submitted 2025-05-18; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: RRMS; cognitive impairment; manual dexterity; bimanual coordination; educational kinesiology program
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Cognitive Dysfunction | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): experimental arm was recieved educational kinesiology program and conventional upper extremity coordination exercises as intervention.Respondents were explained about the Educational kinesiology program.by the therapist. The exercise program was given three times weekly for four weeks. Duration of the session was15 min ), the patients did 5 exercises, each exercise was done for 3 minutes,when patient felt fatigue during performing the exercise he or she stopped then continued after relaxation till reaching 3 min for each one . All exercises were done from sitting position.
  Interventions: Other: educational kinesiology training program intervention for study group; Other: conventional upper extremities coordination training for both arms experimental and comparator (study and control) groups
- control group (Active Comparator): received conventional physical therapy program in form of upper extremities coordination training
  Interventions: Other: conventional upper extremities coordination training for both arms experimental and comparator (study and control) groups

INTERVENTIONS:
Other: educational kinesiology training program intervention for study group — The Educational kinesiology program were included : (Cross crawl) Sit or stand and with the right-hand elbow touch the left knee and vice versa. (The owl) Bring one hand up to the opposite shoulder and hold a pinch around the trapezius muscle between the neck and shoulder. the thumb should be on one side of the muscle and the other fingers clasping around the other side. Turn the head to the same side as thehand is gripping and take a deep breath. Slowly exhale as bringing the head gently around to the other side. Repeat this movement one more time. (The arm activation) Hold one arm next to the ear. Exhale gently while activating the muscles by pushing the arm against the other hand in four directions (front, back, in and away). (The Energizer) Place the head on the desk in front exhale and inhale while coming up and try to hyperextend the neck carefully. (cook's hook-up) put the left ankle over your right knee. Next, hook the right hand around the left ankle.
  Other Names: brain gym exercises
  Arms: study group
Other: conventional upper extremities coordination training for both arms experimental and comparator (study and control) groups — Bimanual coordination,Hand-arm coordination ,Drinking & Strength training

SUMMARY:
the purpose of this study was to evaluate the usefulness of educational kinesiology program to improve cognitive impairement, manual dexterity and bimanual coordination in patients with relapsing remitting multiple sclerosis. the study evaluated some domain of cognition as (attention & concentration, figural memory, reaction behavior and logical reasoning) manual dexterity and bimanual coordination were also evaluated of individuals with multiple sclerosis who went through the traditional as compared to others who used educational kinesiology training as part of their therapy.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic non-curative immune inflammatory demyelinating disease mainly affects the Central Nervous System. Cognitive deficits are common in MS and affect patients at all stages of the disease-including the early stage. There was a negative correlation between the employment of MS patients and their cognitive impairment assessed by information processing speed, memory, and executive function. Currently, the recommended treatments for cognitive dysfunction and depression in people with MS are cognitive retraining and cognitive behavioural therapy, respectively. Both of these approaches are time-consuming and are often unavailable away from major treatment centres. The common clinical signs of the disease include motor and sensory deficits, cerebellar symptoms, fatigue, and/or vision problems, which can impact manipulative dexterity in 76% of the population with MS. Often, patients also present bilateral impairments.Educational kinesiology program is the original 26 movements. The movements which are naturally done during the first years of life when learning coordinated the eyes, ears, hands and whole body are recalled by these activities. The principle behind Educational kinesiology program is that moving with intention leads to optimal learning. Educational kinesiology program has a beneficial effect on cognitive function and combines movement of the feet, hands in the optimization of left and right brain functions so as to improve cognitive function that were damaged or decrease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 18-50 years.
* Patients with relapsing remitting MS (RRMS).
* EDSS scores for (RRMS) is ranging from 2.5 to 5.5 with a pyramid function score less than 2.
* Gave their oral and written consent to participate in the training.
* Adequate vision and hearing for completion of the study protocol, as indicated by the ability to follow written and oral instructions during screening.
* Stable medical condition.

Exclusion Criteria:

* Patients with communication problems.
* Patients with a history of previous neurologic diseases or disorders.
* Patients with other types of MS.
* In co-operative patients.
* Unhealed fracture, contracture, pressure sores that might interfere with training.
* Untreated psychiatric disorders or ongoing drug abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
cognition | baseline assessment and after 12 sessions of educational kinesiology program training and conventional upper extremity coordination exercise training 3 sessions per week for 4 weaks
  the rate of improvement in cognition assessed by Rehacom system V 6.10.2.0 software.

SECONDARY OUTCOMES:
manual dexterity and bimanual coordination | baseline assessment and after 12 sessions of educational kinesiology training and conventional upper extremities coordination exercises training 3 sessions per week for 4 weaks
  manual dexterity and bimanual coordination were assessed by purdue pegboard test model 32107 for purdue pegboard model 32020. assessed the rate of improvement in manual dexterity and bimanual coordination.

CONTACTS AND LOCATIONS:
Overall Officials: eman s fayez, doctorate, Study Director
Locations (1):
- Faculty of Physicaltherapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alharthi HM, Almurdi MM. Association between cognitive impairment and motor dysfunction among patients with multiple sclerosis: a cross-sectional study. Eur J Med Res. 2023 Mar 2;28(1):110. doi: 10.1186/s40001-023-01079-6. PMID 36864515
- [Background] Lyle KB, Dombroski BA, Faul L, Hopkins RF, Naaz F, Switala AE, Depue BE. Bimanual coordination positively predicts episodic memory: A combined behavioral and MRI investigation. Brain Cogn. 2017 Nov;118:71-79. doi: 10.1016/j.bandc.2017.07.009. Epub 2017 Aug 9. PMID 28800429